CLINICAL TRIAL: NCT06766383
Title: Feasibility Study of Using GPT for History-taking Training in Medical Education
Brief Title: Simulated Patient and AI-based Roleplay for History-taking
Acronym: SPAR-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: zhen wang (Other)
Responsible Party: Sponsor-Investigator, zhen wang, physician, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GPT for history-taking Trainin; 2023jyxm1150 (Other Grant/Funding Number: 2023 Anhui Province Quality Engineering Project)
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: History-taking Training; GPT; Medical Education
Keywords: History-taking Training; Artificial Intelligence; Medical Education; GPT Simulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): using GPT-simulated patients
  Interventions: Behavioral: GPT-simulated patients
- control group (Active Comparator): using traditional role-playing
  Interventions: Behavioral: traditional role-playing

INTERVENTIONS:
Behavioral: GPT-simulated patients — GPT-simulated patients
  Arms: intervention group
Behavioral: traditional role-playing — traditional role-playing
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate whether AI-based simulated patient training can improve clinical reasoning and history-taking skills in medical students. The main questions it aims to answer is:

Does GPT-based simulated patient training improve medical students' history-taking skills compared to traditional role-playing methods?

Participants will:

Participants in the intervention group perform medical history-taking conversations with an AI-simulated patient. Receive AI-generated structured feedback on their performance. The control group participated in role-playing exercises with instructors who acted as patients, receiving feedback after each session. Complete standardized assessments to evaluate clinical reasoning and decision-making skills.

ELIGIBILITY:
Inclusion Criteria:Medical education enrollment:

Students enrolled in a medical or health-related professional program.

Clinical coursework completion:

Students who have completed basic clinical coursework, including foundational topics in patient communication and clinical reasoning.

Age group:

Participants aged 18-30 years to reflect typical medical student demographics.

Language proficiency:

Adequate proficiency in the language used for the study (e.g., English) to effectively interact with the AI-simulated patient and understand feedback.

Willingness and availability:

Students who provide informed consent and are willing to participate in all required study activities, including training sessions and assessments.

Access to technology:

Ability to access and use the necessary technology, such as a computer and internet connection, to complete the simulated patient interactions.

-

Exclusion Criteria:Non-medical background:

Students not enrolled in medical or related health professions programs. Students in early years of study who have not completed basic clinical coursework.

Technical limitations:

Inability to access or use the required technology (e.g., computer or online platforms).

Time constraints:

Inability to complete all required training and assessments within the study timeline.

Language barriers:

Insufficient proficiency in the language used for the study (e.g., English) to effectively communicate or understand the simulated patient interactions.

Health-related factors:

Conditions that may impair participation, such as significant hearing or vision impairment, or severe psychological conditions.

Prior participation in similar studies:

Students who have already participated in studies involving similar AI-based simulated patient training or feedback.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
structured clinical examination to measure students' abilities in history taking | From enrollment to the end of treatment at 4 weeks
  Pre and Post Training: This primary endpoint measures improvements in students' clinical skills using a structured clinical examination conducted both before and after the training. The total score is out of 100 points, aggregated from four components:
  History Collection (30 points): Assesses the level of detail in the chief complaint and symptoms (10 points), the ability to understand and identify patient information (10 points), and the appropriateness and logic of follow-up questions (10 points).
  Clinical Reasoning (30 points): Evaluates the thoroughness of diagnostic thinking (15 points) and efficiency in processing information and forming clinical judgments (15 points).
  Communication Skills (20 points): Includes interaction with patients (10 points) and clarity of information delivery (10 points).
  Professional Behavior (20 points): Measures adherence to clinical procedural norms (10 points) and professional attitude towards patients (1

SECONDARY OUTCOMES:
Training Feedback Assessment | From enrollment to the end of treatment at 4 weeks
  Training Feedback Assessment Measurement Tool: Structured Questionnaire on a 5-point Likert scale.
  Components Assessed:
  * Post-class self-directed learning.
  * Enthusiasm for learning.
  * Communication and feedback skills.
  * Expressiveness.
  * Interview logical reasoning ability.
  * Anxiety levels during the interview process. Description: This secondary endpoint collects feedback on the training methods' effectiveness through a structured questionnaire. Each aspect is rated on a 5-point Likert scale, where 1 indicates 'strongly disagree' and 5 indicates 'strongly agree'.
Student Satisfaction Survey | From enrollment to the end of treatment at 4 weeks
  Measurement Tool: Satisfaction Questionnaire on a 5-point Likert scale.
  Components Assessed:
  * Diversity of diseases encountered during training.
  * Naturalness of patient interaction.
  * Usability of the training methods.
  * Likelihood of recommending the training to peers. Description: This secondary endpoint evaluates student satisfaction concerning various aspects of the training experience. The questionnaire assesses each factor on a 5-point Likert scale, where 1 is 'very dissatisfied' and 5 is 'very satisfied'.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Z, Fan TT, Li ML, Zhu NJ, Wang XC. Feasibility study of using GPT for history-taking training in medical education: a randomized clinical trial. BMC Med Educ. 2025 Jul 10;25(1):1030. doi: 10.1186/s12909-025-07614-9. PMID 40640776